CLINICAL TRIAL: NCT01618812
Title: Calcaneal Neck Lengthening Osteotomy - Allogen Bone Graft Material Versus a Hydroxyapatite / β- Tricalcium Phosphate Bone Substitute
Brief Title: Calcaneal Neck Lengthening Osteotomy in Children With Artificial Bone Graft
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-20090162
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Pes Plano Valgus; Flatfeet
Keywords: Artificial bone graft; Hydroxyapatite; Children; Osteotomy; Pes plano valgus; Flatfeet
MeSH Terms: conditions — Flatfoot | interventions — Durapatite

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pes plano valgus: Children with painful flatfeet
  Interventions: Procedure: Lateral lengthening osteotomy of calcaneus

INTERVENTIONS:
Procedure: Lateral lengthening osteotomy of calcaneus — Use of artificial bone graft
  Other Names: Hydroxyapatite

SUMMARY:
In a group of children with severe and painful flatfeet lengthening procedures of calcaneus can be indicated. In this study the investigators use an artificial bone graft technique to avoid removing bone graft from the iliac crest.

DETAILED DESCRIPTION:
The aim is to study the clinical and radiological effects of calcaneal lengthening with either autogen bonegraft or a HA-βTCP graft material in a group of children with planovalgus. The hypothesis is that it is possible to achieve a stabile osteotomy with HA-βTCP graft material equal to the use of autogen bonegraft thus avoiding the need to obtaining iliac crest graft material at growing children.

ELIGIBILITY:
Inclusion Criteria:

* pain
* gait disturbance

Exclusion Criteria:

* post traumatic conditions

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: • children with planovalgus deformity referred to Dept. of Children's Orthopaedics, Dept of Orthopaedic Surgery E, Aarhus University Hospital from June 2009 until January 2012.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Healing of osteotomy | 104 weeks
  Will be followed with repeated clinical examinations until healing

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gottliebsen, PhD-student, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark